CLINICAL TRIAL: NCT02007915
Title: The Use of Bisphosphonates in the Treatment of Avascular Necrosis of the Femoral Head
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decision
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, James Wright, Surgeon-in-Chief & Chief of Perioperative Services, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000009396
Record Dates: First submitted 2013-12-02; First posted 2013-12-11 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Femoral Head Avascular Necrosis
Keywords: Adolescent; Avascular Necrosis; Bisphosphonates; Pamidronate
MeSH Terms: conditions — Femur Head Necrosis; Osteonecrosis | interventions — Pamidronate

ARMS (1):
- Pamidronate Disodium (Experimental)
  Interventions: Drug: Pamidronate Disodium

INTERVENTIONS:
Drug: Pamidronate Disodium — Pamidronate will be given intravenously over one hour, one day per month for three out of every four months. The initial dose is 0.5mg/kg and subsequent doses are 1mg/kg. Infusions will continue for at least one year with a second year possibly recommended by the surgeon from data on the x-ray and bone scan.
  Other Names: Pamidronate Disodium DIN: 002244550

SUMMARY:
To determine the safety and effectiveness of pamidronate in patients with radiographically proven avascular necrosis which are the result of unstable (acute) slipped capital femoral epiphysis, traumatic proximal femur fractures, traumatic hip dislocations, or idiopathic in nature.

DETAILED DESCRIPTION:
Avascular necrosis of the femoral head and collapse is a devastating condition in the pediatric patient population leading to degenerative arthritis and significant disability. Bisphosphonate therapy has been shown to be effective in the treatment of adults with avascular necrosis of the femoral head. For children and adolescents however, there is currently no effective treatment that prevents collapse of the femoral head. Some patients with proven avascular necrosis of the femoral epiphysis are treated with bisphosphonates (intravenous pamidronate) at the The Hospital for Sick Children. The main aim of this study is to prospectively collect data on HSC patients receiving bisphosphonate treatment and thereby report the effectiveness of this treatment in the prevention of femoral head collapse.

ELIGIBILITY:
Inclusion Criteria:

Patients between the ages of 10 and 18 with:

* unstable slipped capital femoral epiphysis (defined as inability to bear weight) or acute slipped capital femoral epiphysis (defined as a separation of the epiphysis from the metaphysis of the proximal femur) who have been pinned either in situ or following reduction,
* traumatic hip dislocations or traumatic proximal femur fractures, or
* "idiopathic" avascular necrosis of the femoral head which includes unknown causes as well as Sickle Cell Disease, post radiation use, post chemotherapy treatment, and post steroid treatment.

Exclusion Criteria:

* Decline to participate in study. (Patients will be still offered this therapy whether or not they wish to be included in the official study protocol. Clinical evaluations, laboratory and imaging tests would be unchanged if they choose to be treated with intravenous pamidronate)
* Significant femoral head collapse - judged radiographically by treating surgeon
* Idiopathic causes under the age of 10.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2011-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Avascular necrosis | 2 years
  Prevention of femoral head collapse and the degree of avascular necrosis following treatment with bisphosphonates as determined clinically and radiographically

SECONDARY OUTCOMES:
Activities Scales for Kids (ASK) | 2 years
  Validated questionnaire (ASK) is used to assess impact of avascular necrosis and femoral head collapse on patient functioning

CONTACTS AND LOCATIONS:
Overall Officials: James Wright, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada